CLINICAL TRIAL: NCT03715881
Title: Scientific Title: Efficacy of Oral Prednisolone and Erythropoietin Injection in Treatment of Acute Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION)
Brief Title: NAION Treatment With Oral Prednisolone and Erythropoietin Injection
Acronym: NAION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Clinical Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 95275
Record Dates: First submitted 2018-06-12; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-06

CONDITIONS: Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION)

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral prednisolone administration (Active Comparator): 50 mg oral prednisolone from the onset of the disease for 1 week, with the dose gradually reduced within 2 weeks and then discontinued
  Interventions: Drug: Oral prednisolone administration 50 mg
- Intravenous Erythropoietin injection (Active Comparator): 2. 1000 units of erythropoietin every 12 hours for three days
  Interventions: Drug: Intravenous Erythropoietin injection

INTERVENTIONS:
Drug: Oral prednisolone administration 50 mg — 50 mg oral prednisolone from the onset of the disease for 1 week, with the dose gradually reduced within 2 weeks and then discontinued
  Arms: Oral prednisolone administration
Drug: Intravenous Erythropoietin injection — 1000 units of erythropoietin every 12 hours for three days
  Arms: Intravenous Erythropoietin injection

SUMMARY:
This randomized double-blind clinical trial is performed on all recent (within the last 5 days) NAION patients referred to hospitals affiliated to the Shahid Beheshti University of Medical Sciences, Iran. The patients will be equally and randomly assigned into two experimental groups and a control group. The first experimental group will receive 1000 units of erythropoietin every 12 hours for three days. The second experimental group will receive 50 mg of oral prednisolone from the onset of the disease for 1 week, with the dose gradually reduced within 2 weeks and then discontinued. In addition, the subjects in the second experimental group will receive 300 mg of ranitidine daily. The third group will receive placebo. Eye examination with color vision, perimetry, and peripapillary optical coherence tomography (to measure the thickness of the retinal nerve fiber layer) will be performed before the intervention, and 1, 3 and 6 months after the intervention. SITA standard visual field testing will be done using the Visual Field Analyzer Humphrey 750 Field (Carl Zeiss, USA). The thickness of the retinal nerve fiber layer will be measured by optical coherence tomography (Cirrus Zeiss Cirrus HD-OCT, Carl Zeiss, USA). The q-q plot and Kolmogorov-Smirnov tests will be performed to test normal distribution of data. Descriptive statistics including frequency, percentages, standard deviation, median and range will be used. Other statistical test including ANOVA, Kruskal-Wallis, Chi-Square, and Fischer's exact tests will be performed. All statistical analyses will be performed in SPSS (version 20) at significance level of 0.05.

ELIGIBILITY:
Inclusion criteria:

- All NAION patients (maximum time of disease occurrence: 5 days) referred to emergency department of Labbafinejad, Torfeh and Imam Hossein hospitals

Exclusion criteria:

1. Glaucoma or any ocular, neurologic or systemic disease affecting the vision
2. Abnormal laboratory test results such as ESR and CRP
3. History of ocular surgery
4. History of receiving medication for NAION
5. Uncontrolled systemic disease such as diabetes or hypertension
6. Contraindications of systemic steroids including active infection, active gastric ulcer, immunosuppression
7. Contraindications of erythropoietin administration, such as polycythemia
8. Unwillingness to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in indices visual acuity compared to normal course of the disease | 6 months after the intervention
  Snellen visual acuity chart
Improvement in indices visual field | 6 months after the intervention
  Mean deviation and pattern standard deviation
Improvement in indices retinal nerve fiber thickness | 6 months after the intervention
  peripapillary Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran